CLINICAL TRIAL: NCT03347734
Title: Randomized Controlled, Double-Blind Trial of Investigation of the Effect of Different Eye Exercises on Hypermetropia in School-age Children
Brief Title: Investigation of the Effect of Different Eye Exercises on Hypermetropia in School-age Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Gülay Aras, Lecturer, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10840098-604.01.01- E.14383
Record Dates: First submitted 2017-11-15; First posted 2017-11-20 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Hyperopia
Keywords: eye exercises; convergence exercise; hyperopia; oculomotor exercise; school-age children
MeSH Terms: conditions — Hyperopia

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Double-Blind Study
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants do not have information about treatment content and groups. He is only aware of exercise therapy applied to him.The ophthalmologist performed evaluations without knowledge of the groups in which the participants were included and of exercise therapy administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Eye Exercises Group (EEG) (Experimental): For the individuals in the group of eye exercises (GEG), 10 repetitive eye exercises protocol was organized as a home program for 6 weeks, twice a day in the morning and evening each day of the week.
  Interventions: Behavioral: Eye exercises group
- Convergence Exercise Group (CEG) (Experimental): For the individuals in the group of convergence exercise, 5 minutes convergence exercise protocol was organized as a home program for 6 weeks, twice a day in the morning and evening each day of the week.
  Interventions: Behavioral: Convergence exercise group
- Oculomotor Exercise Group (OMEG) (Experimental): For the individuals in the group of oculomotor exercise, 10 repetitive, four different oculomotor exercise protocols with eye stabilization were organized as home programs for 6 weeks, twice a day in the morning and evening each day of the week.
  Interventions: Behavioral: Oculomotor Exercise Group (OMEG)

INTERVENTIONS:
Behavioral: Eye exercises group — * 20 times hot water, 20 times cold water washing face in the morning and evening.
  * Palming; 2 hands are rubbed together and warmed up, and the eyes are closed, and 8 digits are drawn with eyes in darkness.
  * 20 blinks
  * Looking at a clock in a circular shape, from 12 to 6, from 6 to 12, from 3 to 9, from 9 to 3, from 2 to 8, from 8 to 2, oblique from 10 to 4, from 4 to 10, and turning the eyes starting from 12 clockwise and counterclockwise. At the end of the exercises, 2-3 minutes of light massage around the eyes and on sunny days, sunbathing was recommended by closing the eyes for 3-5 minutes and swinging to the left and right.
  Arms: Eye Exercises Group (EEG)
Behavioral: Convergence exercise group — * Close eyes for 15 s,
  * Focus on a point 1 to 1.5 ft away for 10 s,
  * Close eyes for 5 s,
  * Focus on a point 20 ft away for 10 s,
  * Close eyes for 5 s,
  * Focus on a point 1 to 1.5 ft away for 10 s,
  * Blink for 5 s,
  * Close eyes for 5 s.
  Arms: Convergence Exercise Group (CEG)
Behavioral: Oculomotor Exercise Group (OMEG) — * The saccadic eye movement exercise included moving the eyes horizontally between two stationary targets while keeping the head still.
  * The smooth pursuit exercise included moving the target horizontally and tracking it with the eyes while keeping the head still.
  * The adaptation X1 exercise included moving the head horizontally while keeping the stationary target in focus.
  * The adaptation X2 exercise included moving the head and target in opposite directions horizontally while tracking the target with the eyes.
  Arms: Oculomotor Exercise Group (OMEG)

SUMMARY:
Hypermetropia in school-aged children is a pathology which is very common and responds to treatments early. No studies have been found in the literature on the efficancy of the hypermetropia treatments with physiotherapy methods. In our study, it was aimed to investigate the effects of different eye exercises on hypermetropia defects in school age children aged 7-17 years and to determine whether exercise protocols have superiority against each other.

DETAILED DESCRIPTION:
60 volunteer school-aged children (30 girls, 30 boys, between 7-17 years of age) were included in our study. 60 participants were randomly divided into three groups: eye exercises, convergence exercises and oculomotor exercise groups. Home exercise protocols were given to all groups for 2 sessions per day for 6 weeks, and regular phone calls were made once a week. Participants were assessed for their hypermetropic grades by autorefractometry, visual acuity by snellen chart, near and sharp visual acuity by activities of daily vision scale, and the health-related quality of life by pediatric quality of life inventory 4.0 version (PEDSQI 4.0) children report.

ELIGIBILITY:
Inclusion Criteria:

* Having hypermetropia eye defects
* Max. having a 1.50 D astigmatism defect
* Using glasses
* Having mental capacity in the level to understand and do exercises
* Not having systemic disease preventing exercise

Exclusion Criteria:

* Having undergone eye surgery
* Having more than 1.50 D astigmatism defect
* Not using glasses

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-06-14 (Actual); Study Completion 2017-10-25 (Actual)

PRIMARY OUTCOMES:
Visual acuity | 6 week
  Snellen chart was used for visual acuity measurement. Snellen "E" was asked to be registered or registered to the device. In visual acuity measurement, individuals were evaluated with their own glasses.

SECONDARY OUTCOMES:
Hypermetropic grade | 6 week
  The refraction defects were measured by autorefractometry, which is frequently used because it provides fast and reliable results in clinic. In the autorefractometry method, the infrared rays sent to the patient's eye are reflected from the retina back to the device and evaluate the refraction defect of the patient
Near and sharp visual acuity | 6 week
  Subscales of activities of daily vision scale, individuals questioning the near vision and sharp vision scores were used. Individuals question the extent to which they can not perform activities because of the difficulty of seeing them, and the degree of difficulty they experience while doing the activity. Points in different categories are summed and converted to a value between 0-100 by the formula. High score gives good visual acuity.
Health-related quality of life | 6 week
  Participants' health-related quality of life was assessed using the Pediatric Quality of Life Inventory Version 4.0 (PedSQI 4.0) Children Report. Score is calculated in 3 areas as total score of scale (SST), total physical health score (FSTP) and total score of psychosocial health (PSTP) which is calculated by calculating emotional, social and school functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Candan Algun, Study Director — Faculty of Health Sciences
Locations (1):
- Istanbul Medipol Universty, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Langer E, Djikic M, Pirson M, Madenci A, Donohue R. Believing is seeing: using mindlessness (mindfully) to improve visual acuity. Psychol Sci. 2010 May;21(5):661-6. doi: 10.1177/0956797610366543. Epub 2010 Mar 19. PMID 20483844
- [Result] Morimoto H, Asai Y, Johnson EG, Lohman EB, Khoo K, Mizutani Y, Mizutani T. Effect of oculo-motor and gaze stability exercises on postural stability and dynamic visual acuity in healthy young adults. Gait Posture. 2011 Apr;33(4):600-3. doi: 10.1016/j.gaitpost.2011.01.016. Epub 2011 Feb 19. PMID 21334899
- [Result] Kang MT, Li SM, Peng X, Li L, Ran A, Meng B, Sun Y, Liu LR, Li H, Millodot M, Wang N. Chinese Eye Exercises and Myopia Development in School Age Children: A Nested Case-control Study. Sci Rep. 2016 Jun 22;6:28531. doi: 10.1038/srep28531. PMID 27329615
- See also: History of eyes exercise — https://en.wikipedia.org/wiki/Eyes_exercise
- Available data/document: Clinical Study Report — https://en.wikipedia.org/wiki/Bates_method